CLINICAL TRIAL: NCT05640323
Title: Prospective Study to Validate the Clinical Accuracy of the Norbert Device to Measure Pulse Rate
Status: Completed | Type: Observational
Sponsor: Norbert Health (Industry)
Collaborators: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: NCP-0002
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy; Arrhythmia
Keywords: medical device; validation; arrhythmia; ECG; pulse rate; Norbert Device; Norbert Health
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Norbert Device — The Norbert Device (ND) is a contactless, noninvasive device that provides measurements of body temperature, oxygen saturation (SpO2), and pulse rate.

SUMMARY:
The study will evaluate the mean average error (MAE) of measuring pulse rate using the Norbert Device (ND) as compared to a reference heart rate measured using an electrocardiogram (ECG).

DETAILED DESCRIPTION:
The study design is to validate the pulse and heart rate accuracy as required per ISO 80601-2-61, Clause 201.12.1.104. The study is a non-randomized, non-blinded single arm design to evaluate the clinical accuracy of the ND's pulse rate measurement compared to a reference heart rate manually measured by observing R-peaks in a standard concurrently recorded ECG from an FDA 510(k)-cleared reference clinical ECG (RCECG). The sponsor will ensure that the study staff enrolls a range of types of arrhythmias including tachycardia, bradycardia, atrial fibrillation, bigeminy, trigeminy, and others.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 or over
* Ability to provide signed informed consent

Exclusion Criteria:

* Pregnant
* Otherwise deemed unsuitable to participate in the study based on judgment of the study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will recruit subjects within an Emergency Department as well as through online internet bulletin boards.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Mean Average Error (MAE) | Up to 1 hour
  MAE will be evaluated by Mean absolute error (MAE) of the pulse rate of the device compared to the heart rate measured from the RCECG.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Newlab, Brooklyn, New York
  - Staten Island University Hospital, Staten Island, New York

IPD SHARING:
Plan to Share IPD: No